CLINICAL TRIAL: NCT01637363
Title: Psychoeducation to Sick-listed Individuals With Mental Health Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 11-2-2-011; 7-11-1347 (Other Grant/Funding Number: Tryg Fonden)
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Stress, Psychological
Keywords: Psychoeducation; Stress; Sickness absence; Psychiatric symptoms; Locus of control; Self reported health
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular treatment (No Intervention): This group is offered regular treatment from the job center i.e. exercise, mindfulness
- Psychoeducation (Experimental): 6 x 2 hours of psychoeducation
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Psychoeducation — 6 x 2 hours of psychoeducation
  Arms: Psychoeducation

SUMMARY:
In Denmark, it is estimated that 35-45% of all sick leave registered citizens are on sick leave due to psychiatric sufferings. Mental health conditions are of great consequence not only to the sick-listed individual but also to his/her family and to society in general and in socioeconomic terms.

The aim of this project is to systematically compare psychoeducation with the various standard offers to sick listed individuals with mental health conditions provided by job centers in four municipalities.

Psychoeducation is employed within the psychiatric healthcare system and is defined as a group based treatment by means of educating participants about psychiatric conditions. In the present project, the employed psychoeducation focuses on psyche and work life, and its purpose is to impart knowledge about psychiatric conditions in order to provide the sick listed individuals with qualifications to understand, and, thereby, improve their own situation. Among others, there will be information about the symptoms of various psychiatric conditions, diagnoses, and treatment options. Furthermore, the participants will learn about specific, useful, cognitive tools in regards to the barriers and difficulties they might experience when reentering the work force and leave sickness absence behind.

The project is designed as a randomized clinical trial in which the participants are offered either 1) psychoeducation as well as the standard offer to sick listed individuals provided by the municipality in which the individual lives or 2) the participants are offered merely the standard offer to sick listed individuals provided by the municipality.

The target group consists of recently sick listed individuals with mental health issues - whether diagnosed or not. The individuals must be inhabitants of the municipalities of Struer, Lemvig, Skive, and Holstebro.

The outcome measure is the determined as the duration of the sickness absence, the severity of the psychiatric condition, self-reported health, and 'locus of control´. These outcome measurements are assessed at baseline and after 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* A score of 5 or more on SCL-8AD

Exclusion Criteria:

* Sick listed due to psychiatric symptoms in a period of 3 months or longer in the last year
* pregnant
* has a flexible job
* receive pension
* not communicating in Danish

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2012-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
length of sickness absence | 6 months after randomization

SECONDARY OUTCOMES:
Locus of control | Baseline, 3 and 6 months after randomization
Self reported health | Baseline, 3 and 6 months after randomization
Psychological symptoms | Baseline, 3 and 6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Hans Jørgen Søgaard, MD, ph.d., Study Chair — Psychiatric Research Unit West, Regional Psychiatric Services; Pernille Pedersen, MHs, Principal Investigator — Psychiatric Research Unit West, Regional Psychiatric Services; Ellen A Nøhr, ph.d., Study Chair — Institute of Clinical Research, University of Southern Denmark; Chris Jensen, ph.d., Study Chair — National Advisory Unit for Occupational Rehabilitation, Rauland, Norway
Locations (1):
- Psychiatric Research Unit West, Regional Psychiatric Services, Herning, Denmark

REFERENCES:
- [Derived] Pedersen P, Sogaard HJ, Labriola M, Nohr EA, Jensen C. Effectiveness of psychoeducation in reducing sickness absence and improving mental health in individuals at risk of having a mental disorder: a randomised controlled trial. BMC Public Health. 2015 Aug 8;15:763. doi: 10.1186/s12889-015-2087-5. PMID 26253219
- [Derived] Pedersen P, Sogaard HJ, Yde BF, Labriola M, Nohr EA, Jensen C. Psychoeducation to facilitate return to work in individuals on sick leave and at risk of having a mental disorder: protocol of a randomised controlled trial. BMC Public Health. 2014 Dec 17;14:1288. doi: 10.1186/1471-2458-14-1288. PMID 25516423